CLINICAL TRIAL: NCT03253029
Title: Use of Branched-chain Amino Acids in Cancer Cachexia
Brief Title: Study of Branched-chain Amino Acids in Cancer Cachexia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of institutional support
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Principal Investigator, Jordan Waypa, Jordan Waypa, FNP-C, Western Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WG2014009
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cancer Cachexia
Keywords: oncology, cancer cachexia, cachexia anorexia,
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): (arm 1) consume five scoops total per day of Pure Encapsulations Branched Chain Amino Acid powder on an outpatient basis (take 2 scoops both in the morning and afternoon and 1 scoop in the evening)
  Interventions: Dietary Supplement: Pure Encapsulations Branched Chain Amino Acid powder
- Control (Placebo Comparator): (arm 2): control group (no BCAAs provided)
  Interventions: Dietary Supplement: control group (no BCAAs provided)

INTERVENTIONS:
Dietary Supplement: Pure Encapsulations Branched Chain Amino Acid powder
  Arms: Treatment
Dietary Supplement: control group (no BCAAs provided)
  Arms: Control

SUMMARY:
Investigate whether supplementation with branched-chain amino acids (BCAAs) has a positive effect on cancer cachexia, as measured by the maintenance or increase in weight and lean body mass (LBM) based on body weight in kilograms (kg) and bioelectrical impedance assessment (BIA).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Eastern Cooperative Oncology Group (ECOG) performance status score < 2 and a life expectancy >3 months
3. Participants must have evaluable disease by RECIST 1.1 criteria17
4. At least four (4) weeks from prior major surgery
5. Participants must be cachectic as defined by the guidelines below18

   * >5% weight loss over the past 6 months (in absence of simple starvation); OR
   * BMI <20 and any degree of weight loss >2%; OR
   * Appendicular skeletal muscle index consistent with sarcopenia (whole body fat-free mass index without bone determined by bioelectrical impedance (men <14.6 kg/m²; women <11.4 kg/m²) and weight loss >2%
6. Participants must be anorexic as defined by reporting one of the following symptoms below3

   * Early satiety
   * Nausea/vomiting
   * Taste alterations
   * Smell alterations
   * Meat aversion

Exclusion Criteria:

1. Patients taking Levadopa
2. Patients with amyotrophic lateral sclerosis (ALS)
3. Patients utilizing a percutaneous gastrostomy tube for drainage
4. Patients unable to consume food or beverage orally
5. Patients on any form of parenteral nutrition which contains BCAA.
6. Serious non-healing wound, ulcer, or burn
7. Patients who are pregnant or lactating
8. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements
9. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Estimated); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Investigate whether supplementation with BCAAs has a positive effect on cancer cachexia, as measured by the maintenance or increase in weight and LBM based on body weight in kg | 12 weeks
  Investigate whether supplementation with branched-chain amino acids (BCAAs) has a positive effect on cancer cachexia, as measured by the maintenance or increase in weight and lean body mass (LBM) based on body weight in kilograms (kg)
Investigate whether supplementation with BCAAs has a positive effect on cancer cachexia, as measured by the maintenance or increase in BIA | 12 weeks
  Investigate whether supplementation with BCAAs has a positive effect on cancer cachexia, as measured by the maintenance or increase in bioelectrical impedance assessment (BIA).

SECONDARY OUTCOMES:
Examine whether supplementation with BCAAs improve appetite and quality of life based on the MD Anderson Symptom Inventory (MDASI). | 12 weeks